CLINICAL TRIAL: NCT01017146
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of Tazarotene Foam, 0.1%, in Subjects With Acne Vulgaris
Brief Title: A Study to Evaluate the Safety and Efficacy of Tazarotene Foam, 0.1%, in Subjects With Common Facial Acne - W0260-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114575
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Acne Vulgaris
Keywords: Ance
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tazarotene foam, 0.1%
  Interventions: Drug: Tazarotene foam
- 2 (Placebo Comparator): Vehicle Foam
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Tazarotene foam — Tazarotene foam once a day application to the face
  Arms: 1
Drug: Vehicle Foam — Vehicle Foam once a day application to the face
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety and efficacy of a new foam formulation of tazarotene in subjects with acne vulgaris.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, vehicle-controlled, parallel-group study comparing tazarotene foam with vehicle foam in subjects with acne vulgaris. Approximately 742 subjects will be enrolled and randomized to 1 of the 2 study product groups in a 1:1 ratio (tazarotene foam: vehicle foam). Subjects will apply tazarotene foam or vehicle foam to the entire face once daily for 12 weeks; study visits will occur at baseline (week 0/day 1) and at weeks 2, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 12 through 45 years, inclusive, who is in good general health.
* An ISGA score of 3 or greater at baseline.
* Lesion counts meeting both of the following criteria:

  1. Between 25 and 50 facial inflammatory lesions and no more than 1 facial nodular lesion (<5mm), with NO cystic lesions.
  2. Between 30 and 125 facial noninflammatory lesions, excluding nasal lesions.
* Regular menstrual cycle prior to study entry for females of childbearing potential.
* Negative urine pregnancy test for females of childbearing potential. • Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses.

Women who are not currently sexually active must agree to use medically accepted method of contraception should they become sexually active while participating in the study. Male subjects and/or their partners must use a medically acceptable form of contraception.

* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* Ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* Use of topical antibiotics on the face within the past 2 weeks.
* Use of systemic antibiotics for acne treatment within the past 4 weeks.
* Concurrent use of medications known to be photosensitizers (eg, thiazides, tetracyclines) because of the possibility of augmented photosensitivity.
* Use of topical corticosteroids on the face within the past 2 weeks or systemic corticosteroids within the past 4 weeks.
* Use of systemic retinoids (eg, isotretinoin) within the past 6 months.
* Treatment with estrogens, androgens, or anti-androgenic agents for 12 weeks or less immediately prior to study enrollment. Subjects that have been treated with these medications for more than 12 consecutive weeks prior to study enrollment are allowed to enroll as long as they do not expect to change the dose or drug, or to discontinue use during the study and it has not been indicated for the treatment of acne vulgaris.
* Use of topical anti-acne medications (eg, benzoyl peroxide, retinoids, or salicylates) within the past 2 weeks.
* Concomitant use of facial products such as: abradants, facials, peels containing glycolic or other acids, masks, washes or soaps.
* Concomitant use of medications that are reported to exacerbate acne (eg, mega-doses of certain vitamins, haloperidol, and immunosuppressants such as cyclosporine) as these may impact efficacy assessments. Multivitamins, iron supplements, and folate are acceptable.
* Facial procedure (eg, blue light, chemical or laser peel, or microdermabrasion) within the past 4 weeks.
* Require or desire excessive or prolonged exposure to ultraviolet light during the study.
* Known hypersensitivity or previous allergic reaction to any of the active components of the study product.
* A significant medical history of or currently immunocompromised.
* Use of any investigational product within the past 4 weeks or currently participating in another clinical study.
* Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.
* Any major illness within 30 days before study enrollment.
* Currently lives in the same household as currently enrolled subjects; is an employee of Stiefel, an investigator, or a CRO involved in the study; or is an immediate family member (eg, partner, offspring, parents) of an employee involved in the study

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 744 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (19):
  - Cherry Creek Research, Inc., Denver, Colorado
  - Cosmetic Medicine & Treatment Research Insttitute, Inc., Miami Beach, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - DermResearch Center of New York, Inc., Stony Brook, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Dermatology Research of Cincinnati, Cincinnati, Ohio
  - Group Health Associates, Cincinnatti, Ohio
  - Haber Dermatology & Cosmetic Surgery, Inc., South Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Dermatology Research Associates, Inc., Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Aurora Advanced Healthcare, Inc. Clinical Research Center, Milwaukee, Wisconsin
- Canada (3):
  - Ultranova Skincare, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Nexus Clinical Research, St. John's

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Feldman SR, Werner CP, Alio Saenz AB. The efficacy and tolerability of tazarotene foam, 0.1%, in the treatment of acne vulgaris in 2 multicenter, randomized, vehicle-controlled, double-blind studies. J Drugs Dermatol. 2013 Apr;12(4):438-46. PMID 23652892
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tazarotene Foam: Tazarotene foam containing 0.1% tazarotene in an emulsion formulation foam vehicle was applied to the face once daily in the early evening for 12 weeks. A sufficient amount of study product was applied to cover the entire face and was gently rubbed into the skin until the study product disappeared. Tazarotene foam was packaged in a 100-gram aluminum can pressurized with a hydrocarbon propellant.
- Vehicle Foam: The matching vehicle foam containing only tazarotene foam vehicle was applied to the face once daily in the early evening for 12 weeks. A sufficient amount of study product was applied to cover the entire face and was gently rubbed into the skin until the study product disappeared. Vehicle foam was packaged in a 100-gram aluminum can pressurized with a hydrocarbon propellant.
Period: Overall Study
Arm/Group | Tazarotene Foam | Vehicle Foam
Started | 372 | 372
Completed | 306 | 333
Not Completed | 66 | 39
Not completed — Adverse Event | 11 | 1
Not completed — Lost to Follow-up | 14 | 14
Not completed — Noncompliance with Study Product | 1 | 1
Not completed — Withdrawal by Subject | 32 | 16
Not completed — Relocation | 0 | 4
Not completed — Pregnancy | 2 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Took Excluded Medication | 2 | 0
Not completed — Did Not Meet Eligibility Criteria | 1 | 2
Not completed — Change in Work Situation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tazarotene Foam | Vehicle Foam | Total
Number analyzed (Participants) | 371 | 372 | 743
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Analysis Set, consisting of all randomized participants who were dispensed study product. One participant was randomized to the tazarotene foam group, but discontinued due to pregnancy and did not receive study product.
  Years
    Years | 18.2 (5.7) | 18.6 (6.4) | 18.4 (6.1)
Gender [Count of Participants; unit: Participants] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Analysis Set, consisting of all randomized participants who were dispensed study product. One participant was randomized to the tazarotene foam group, but discontinued due to pregnancy and did not receive study product.
  Participants
    Female | 182 | 192 | 374
    Male | 189 | 180 | 369
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristics were collected in members of the Intent-to-Treat (ITT) Analysis Set, consisting of all randomized participants who were dispensed study product. One participant was randomized to the tazarotene foam group, but discontinued due to pregnancy and did not receive study product.
  participants
    American Indian or Alaska Native | 12 | 3 | 15
    Asian | 11 | 4 | 15
    Black | 53 | 50 | 103
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    White | 285 | 307 | 592
    Mixed Race | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Lesion Counts (LCs) From Baseline to Week 12
Description: LC: count of all inflammatory lesions (ILs, i.e., papules, pustules, and nodules) and non-inflammatory lesions (NILs, i.e., open and closed comedones) at Baseline and at Week 12. Total lesions (TLs) were calculated as the sum of ILs and NILs. LC was confined to the face (including forehead, nose, checks, and chin). Change from Baseline at Week 12 was calculated as the value at Week 12 minus the value at Baseline.
Time Frame: Baseline (Week 0/Day 1) and Week 12
Population: Intent-to-Treat (ITT) Analysis Set: all randomized participants who were dispensed study product. Calculation was based on the last observation carried forward (LOCF) imputation method for missing data, in which missing final values of the outcome variable are replaced by the last known value before the participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: lesion counts
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
lesion counts
  ILs | -18.0 (11.01) | -14.1 (12.37)
  NILs | -27.9 (21.65) | -16.7 (21.72)
  TLs | -45.8 (27.89) | -30.8 (26.68)
Statistical Analysis 1: Comparison: Tazarotene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value indicates treatment differences between tazarotene foam and vehicle foam for ILs
Statistical Analysis 2: Comparison: Tazarotene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value indicates treatment differences between tazarotene foam and vehicle foam for NILs
Statistical Analysis 3: Comparison: Tazarotene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value indicates treatment differences between tazarotene foam and vehicle foam for TLs

2. Primary Outcome: Number of Participants With a Minimum 2-grade (G) Improvement in the Investigator Static Global Assessment (ISGA) Score From Baseline at Week 12
Description: Investigators evaluated the acne severity (S) of the participants' face using the ISGA scale, ranging from 0 to 5: 0=clear skin with no ILs or NILs; 1=almost clear: rare NIL with no more than rare papules; 2=mild S: >G 1, some NILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate S: >G 2, up to many NILs and may have some ILs, but no more than one small NL; 4=severe: greater than G 3, up to many NILs and ILs, but no more than a few NLs; 5=very severe: many NILs and ILs and more than a few NLs, may have cystic lesions.
Time Frame: Baseline (Week 0/Day 1) and Week 12
Population: ITT Analysis Set
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
participants | 132 | 89
Statistical Analysis 1: Comparison: Tazarotene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage of participants = 35.6, 95% CI 2-sided [30.7 to 40.5] — The estimated value represents the percentage of participants receiving tazarotene foam with a minimum 2 G improvement in the ISGA score from Baseline at Week 12
Statistical Analysis 2: Comparison: Vehicle Foam; Test type: Superiority or Other; Percentage of participants = 23.9, 95% CI 2-sided [19.6 to 28.3] — The estimated value represents the percentage of participants receiving vehicle foam with a minimum 2 G improvement in the ISGA score from Baseline at Week 12

3. Primary Outcome: Number of Participants With an ISGA Score of 0 or 1 at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: ITT Analysis Set. Missing values were imputed using the LOCF method.
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
participants | 107 | 60
Statistical Analysis 1: Comparison: Tazarotene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage of participants = 28.8, 95% CI 2-sided [24.2 to 33.5] — The estimated value represents the percentage of participants receiving tazarotene foam with an ISGA score of 0 or 1 at Week 12
Statistical Analysis 2: Comparison: Vehicle Foam; Test type: Superiority or Other; Percentage of participants = 16.1, 95% CI 2-sided [12.4 to 19.9] — The estimated value represents the percentage of participants receiving vehicle foam with an ISGA score of 0 or 1 at Week 12

4. Secondary Outcome: Percent Change in LC From Baseline at Weeks 2, 4, 8, and 12
Description: LC: count of all ILs (i.e., papules, pustules, and nodules) and NILs (i.e., open and closed comedones) at Baseline and at Week 12. TLs were calculated as the sum of ILs and NILs. LC was confined to the face (including forehead, nose, checks, and chin). Percent change from Baseline in LC at Weeks 2, 4, 8, and12 was calculated as the (Week 2/4/8/12 value minus the baseline value divided by baseline value) x 100.
Time Frame: Baseline (Week 0/Day 1); Weeks 2, 4, 8, and 12
Population: ITT Analysis Set. The LOCF imputation method was used for missing data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
percent change
  ILs, Week 2 | -18.2 (35.84) | -20.9 (33.64)
  ILs, Week 4 | -33.0 (32.75) | -24.8 (34.42)
  ILs, Week 8 | -50.1 (31.53) | -42.1 (38.62)
  ILs, Week 12 | -57.5 (33.39) | -45.2 (38.64)
  NILs, Week 2 | -24.5 (26.21) | -16.6 (28.64)
  NILs, Week 4 | -36.6 (28.59) | -25.0 (32.45)
  NILs, Week 8 | -48.7 (29.20) | -30.6 (36.64)
  NILs, Week 12 | -55.1 (30.88) | -34.3 (42.56)
  TLs, Week 2 | -22.5 (23.39) | -18.8 (22.21)
  TLs, Week 4 | -35.3 (25.41) | -29.3 (26.98)
  TLs, Week 8 | -49.5 (26.2) | -35.6 (31.16)
  TLs, Week 12 | -56.3 (28.52) | -39.0 (34.40)

5. Secondary Outcome: Absolute Change From Baseline in LC at Weeks 2, 4, and 8
Description: LC: count of all ILs (i.e., papules, pustules, and nodules) and NILs (i.e., open and closed comedones) at Baseline and at Week 12. TLs were calculated as the sum of ILs and NILs. LC was confined to the face (including forehead, nose, checks, and chin). Change from Baseline at Week 12 was calculated as the value at Week 12 minus the value at baseline. Calculation was based on last observation carried forward (LOCF) imputation method for missing data.
Time Frame: Baseline (Week 0/Day 1); Weeks 2, 4, and 8
Population: ITT Analysis Set. Calculation was based on the LOCF imputation method for missing data.
Measure: Mean (Standard Deviation); unit: lesion counts
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
lesion counts
  ILs, Week 2 | -5.5 (11.54) | -6.5 (11.98)
  ILs, Week 4 | -10.1 (10.44) | -10.9 (11.74)
  ILs, Week 8 | -15.6 (10.40) | -13.2 (12.71)
  NILs, Week 2 | -12.6 (15.72) | -8.6 (16.22)
  NILs, Week 4 | -18.2 (17.70) | -12.2 (18.41)
  NILs, Week 8 | -24.6 (19.64) | -14.8 (21.63)
  TLs, Week 2 | -18.1 (20.22) | -15.1 (18.80)
  TLs, Week 4 | -28.3 (22.77) | -23.1 (23.30)
  TLs, Week 8 | -40.1 (24.67) | -27.9 (28.09)

6. Secondary Outcome: Time to a 50 Percent Reduction in Total Lesion Counts (TLC)
Description: Time to a 50 percent reduction in TLC (sum of ILs and NILs) was the time difference between Baseline and the time to 50 percent reduction in LC. Participants who did not have a >=50 percent reduction from Baseline in TLC during the study were censored at their last visit date.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: ITT Analysis Set: only those participants with a >=50 percent reduction from Baseline in TLC were evaluated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 273 | 197
days | 57 [57 to 58] | 85 [80 to 86]

7. Secondary Outcome: Number of Participants With a Minimum 2-grade Improvement in ISGA Score at Weeks 2, 4, and 8
Description: as for outcome 2
Time Frame: Baseline (Week 0/Day 1); Weeks 2, 4, and 8
Population: ITT Analysis Set
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
participants
  Week 2 | 10 | 11
  Week 4 | 23 | 29
  Week 8 | 64 | 44

8. Secondary Outcome: Number of Participants With an ISGA Score of 0 or 1 at Weeks 2, 4, and 8
Description: as for outcome 2
Time Frame: Weeks 2, 4, and 8
Population: ITT Analysis Set. Missing values were imputed using the LOCF method.
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
participants
  Week 2 | 4 | 1
  Week 4 | 12 | 7
  Week 8 | 40 | 22

9. Secondary Outcome: Number of Participants With a Subject's Global Assessment (SGA) Score of 0 or 1 at Weeks 2, 4, 8, and 12
Description: An SGA of the facial skin, excluding the scalp, was performed by participants using a rating scale of 0 to 4: 0=face is basically free of acne, with only an occasional blackhead (Bh) and/or whitehead (Wh); 1=face has several Bhs and/or Whs and small pimples (P), but there are no tender deep-seated bumps or cysts (DSBCs); 2=face has several to many Bhs and/or Whs and small- to medium-sized P, and may have one DSBC; 3=face has many Bhs and/or Whs, many medium- to large-sized P, and perhaps a few DSBCs; 4=face has Bhs and/or Whs, and several to many medium- to large-sized Ps and DSBCs dominate.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Analysis Set
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 371 | 372
participants
  Week 2 | 104 | 1
  Week 4 | 143 | 130
  Week 8 | 187 | 165
  Week 12 | 220 | 180

10. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Baseline at Weeks 2, 4, 8, and 12 in Participants 17 Years of Age or Older
Description: The DLQI was used to measure how much the participants' skin problem had affected their life over the last week. The DLQI total score ranges from 0 to 30: 0-1=no effect at all on the participant's life; 2-5=small effect on the participant's life; 6-10=moderate effect on the participant's life; 11-20=very large effect on the participant's life; 21-30=extremely large effect on the participant's life. A lower score on the DLQI indicates increased quality of life; therefore, negative changes from Baseline indicate improvements.
Time Frame: Baseline (Week 0/Day 1); Weeks 2, 4, 8, and 12
Population: ITT Analysis Set: only those participants 17 years of age or older and whose DLQI scores were calculated at Baseline and at Weeks 2, 4, 8, or 12 were evaluated for change in DLQI score at the respective week.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 171 | 165
Scores on a scale
  Week 2, n=171,165 | -0.1 (4.98) | -2.1 (3.68)
  Week 4, n=166, 167 | -1.9 (4.60) | -2.5 (3.85)
  Week 8, n=160, 155 | -2.9 (4.86) | -2.7 (4.40)
  Week 12, n=154, 155 | -3.6 (5.22) | -3.1 (4.31)

11. Secondary Outcome: Change in Children's Dermatology Life Quality Index (CDLQI) From Baseline at Week 2, 4, 8 and 12 in Participant's With 16 Years Old or Younger
Description: The CDLQI was used to measure how much the participants' skin problem had affected their life over the last week. The CDLQI total score ranges from 0 to 30: 0-1=no effect at all on the participant's life; 2-6=small effect on the participant's life; 7-12=moderate effect on the participant's life; 13-18=very large effect on the participant's life; 19-30=extremely large effect on the participant's life. A lower score on the CDLQI indicates increased quality of life; therefore, negative changes from Baseline indicate improvements.
Time Frame: Baseline (Week 0/Day 1); Weeks 2, 4, 8, and 12
Population: ITT Analysis Set: only those participants 16 years of age or younger and whose CDLQI scores were calculated at Baseline and at Weeks 2, 4, 8, or 12 were evaluated for change in DLQI score at the respective week.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 162 | 179
scores on a scale
  Week 2, n=162,179 | 1.1 (4.16) | -1.4 (3.21)
  Week 4, n=153, 180 | -0.6 (3.45) | -1.4 (3.23)
  Week 8, n=148, 171 | -1.2 (3.53) | -1.9 (3.11)
  Week 12, n=146, 169 | -1.7 (4.09) | -2.0 (3.46)

12. Secondary Outcome: Number of Participants With the Indicated Local Tolerability Assessment for Erythema as Evaluated by the Investigator
Description: Erythema is a skin condition characterized by redness or rash. Local tolerability assessments were performed by the Investigator at each study visit and were graded based on severity as G0 to G4: G0=absent (no redness); G1=slight (faint red or pink coloration, barely perceptible); G2=mild (light red or pink coloration); G3=moderate (medium red coloration); G4=severe (beet red coloration). Maximum During Treatment is defined as the maximum severity of erythema reported at any time during treatment.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: All Randomized Participants: all participants who were randomized in the study
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 372 | 372
participants
  Baseline, G0 | 250 | 242
  Baseline, G1 | 69 | 99
  Baseline, G2 | 45 | 24
  Baseline, G3 | 7 | 7
  Baseline, G4 | 0 | 0
  Baseline, Missing G | 1 | 0
  Maximum During Treatment (MDT), G0 | 81 | 133
  MDT, G1 | 99 | 152
  MDT, G2 | 115 | 64
  MDT, G3 | 64 | 13
  MDT, G4 | 3 | 0
  MDT, Missing G | 10 | 10
  Week 12, G0 | 159 | 216
  Week 12, G1 | 83 | 87
  Week 12, G2 | 50 | 24
  Week 12, G3 | 11 | 3
  Week 12, G4 | 1 | 0
  Week 12, Missing G | 68 | 42

13. Secondary Outcome: Number of Participants With the Indicated Local Tolerability Assessment for Drying as Evaluated by the Investigator
Description: Dryness: skin epidermis that lacks moisture/sebum. Local tolerability assessments were performed by the Investigator at each study visit and were graded based on severity as G0 to G4. G0=absent (none); G1=slight (barely perceptible dryness with no flakes or fissure formation); G2=mild (easily perceptible dryness with no flakes or fissure formation); G3=moderate (easily noted dryness and flakes but no fissure formation); G4=severe (easily noted dryness with flakes and fissure formation). Maximum During Treatment is defined as the maximum severity of drying reported at any time during treatment.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: All Randomized Participants
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 372 | 372
participants
  Baseline, G0 | 329 | 327
  Baseline, G1 | 34 | 36
  Baseline, G2 | 6 | 9
  Baseline, G3 | 2 | 0
  Baseline, G4 | 0 | 0
  Baseline, Missing G | 1 | 0
  MDT, G0 | 96 | 222
  MDT, G1 | 101 | 102
  MDT, G2 | 90 | 36
  MDT, G3 | 72 | 2
  MDT, G4 | 3 | 0
  MDT, Missing G | 10 | 10
  Week 12, G0 | 208 | 292
  Week 12, G1 | 67 | 33
  Week 12, G2 | 22 | 5
  Week 12, G3 | 7 | 0
  Week 12, G4 | 0 | 0
  Week 12, Missing G | 68 | 42

14. Secondary Outcome: Number of Participants With the Indicated Local Tolerability Assessment for Peeling as Evaluated by the Investigator
Description: Peeling skin: damage to and loss of the upper layer of skin (epidermis). Local tolerability assessments for peeling were performed by the Investigator at each study visit and were graded based on severity as G0 to G4: G0=absent (no peeling); G1=slight (mild localized peeling); G2=mild (mild and diffuse peeling); G3=moderate (moderate and diffuse peeling); G4=severe (moderate to prominent, dense peeling). Maximum During Treatment is defined as the maximum severity of peeling reported at any time during treatment.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: All Randomized Participants
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 372 | 372
participants
  Baseline, G0 | 344 | 339
  Baseline, G1 | 22 | 29
  Baseline, G2 | 5 | 4
  Baseline, G3 | 0 | 0
  Baseline, G4 | 0 | 0
  Baseline, Missing G | 1 | 0
  MDT, G0 | 112 | 256
  MDT, G1 | 104 | 76
  MDT, G2 | 87 | 28
  MDT, G3 | 51 | 2
  MDT, G4 | 8 | 0
  MDT, Missing G | 10 | 10
  Week 12, G0 | 221 | 300
  Week 12, G1 | 57 | 25
  Week 12, G2 | 16 | 5
  Week 12, G3 | 10 | 0
  Week 12, G4 | 0 | 0
  Week 12, Missing G | 68 | 42

15. Secondary Outcome: Number of Participants With the Indicated Local Tolerability Assessment for Itching as Evaluated by the Participants
Description: Itching is a sensation that causes the desire or reflex to scratch. Local tolerability assessments for itching were performed by the participant at each study visit and were graded based on severity as G0 to G3. G0=none; G1=slight; G2=moderate; G3=strong. Maximum During Treatment is defined as the maximum severity of itching reported at any time during treatment.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: All Randomized Participants
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 372 | 372
participants
  Baseline, G0 | 237 | 229
  Baseline, G1 | 104 | 109
  Baseline, G2 | 26 | 30
  Baseline, G3 | 3 | 4
  Baseline, Missing G | 2 | 0
  MDT, G0 | 68 | 126
  MDT, G1 | 164 | 182
  MDT, G2 | 92 | 48
  MDT, G3 | 38 | 6
  MDT, Missing G | 10 | 10
  Week 12, G0 | 174 | 216
  Week 12, G1 | 111 | 96
  Week 12, G2 | 17 | 16
  Week 12, G3 | 2 | 2
  Week 12, Missing G | 68 | 42

16. Secondary Outcome: Number of Participants With the Indicated Local Tolerability Assessment for Burning/Stinging as Evaluated by the Participants
Description: Burning/stinging is a pain and burning sensation. Local tolerability assessments were performed by the participant at each study visit based on severity as G0 to G3: G0=none; G1=slight; G2=moderate; G3=strong. Maximum During Treatment is defined as the maximum severity of burning/stinging reported at any time during treatment.
Time Frame: Baseline (Week 0/Day 1) to Week 12
Population: All Randomized Participants
Measure: Number; unit: participants
Arm/Group | Tazarotene Foam | Vehicle Foam
Number analyzed (Participants) | 372 | 372
participants
  Baseline, G0 | 307 | 291
  Baseline, G1 | 34 | 64
  Baseline, G2 | 26 | 15
  Baseline, G3 | 3 | 2
  Baseline, Missing G | 2 | 0
  MDT, G0 | 52 | 137
  MDT, G1 | 101 | 159
  MDT, G2 | 122 | 55
  MDT, G3 | 87 | 11
  MDT, Missing G | 10 | 10
  Week 12, G0 | 179 | 222
  Week 12, G1 | 94 | 94
  Week 12, G2 | 24 | 13
  Week 12, G3 | 7 | 1
  Week 12, Missing G | 68 | 42

ADVERSE EVENTS:
Arm/Group | Tazarotene Foam | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 1/371 | 1/372
Other Adverse Events (participants affected / at risk) | 88/371 | 17/372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazarotene Foam (N=371) | Vehicle Foam (N=372)
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Adjustment disorder with mixed disturbance of emotion, condu (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tazarotene Foam (N=371) | Vehicle Foam (N=372)
Application Site Dryness (General disorders) | 22 | 2
Application Site Irritation (General disorders) | 66 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.